CLINICAL TRIAL: NCT05602753
Title: Carbon Monoxide Breath Testing Prior to Total Joint Arthroplasty to Ascertain Smoking and Aid in Encouraging Smoking Cessation
Brief Title: Smoking Cessation Study
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Responsible Party: Principal Investigator, Adam Hart, Principal Investigator, Staff Orthopaedic Surgeon, McGill University Health Centre/Research Institute of the McGill University Health Centre
Other Study IDs: 2020-6424
Record Dates: First submitted 2022-10-27; First posted 2022-11-02 (Actual); Last update posted 2022-11-04 (Actual); Status verified 2022-11

CONDITIONS: Smoking Cessation; Arthropathy
MeSH Terms: conditions — Smoking Cessation; Joint Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Smokers: All patients who participate in the study will complete the smoking history questionnaire and the carbon monoxide breath test. All patients with positive carbon monoxide breath test indicative of active nicotine exposure will be provided a structured smoking cessation program that includes information, counseling from their surgeon, or a trained health care professional and referral to a smoking cessation program.
  Interventions: Behavioral: Lifestyle Counseling
- Non-Smokers: Subjects who self-declared as non-smokers
- Declared non-smokers with elevated Co2: subjects who self-declared as non-smokers but who tested positive for elevated Co2,

INTERVENTIONS:
Behavioral: Lifestyle Counseling — Referring to Stop smoking hotline, given pamphlets to encourage quitting smoking, pharmacy guidance, and possible referral to smoking cessation clinic.
  Groups: Smokers

SUMMARY:
The primary outcome of this study is to determine the true incidence of smokers among patients undergoing joint replacement and secondly, what percent are able to quit smoking before surgery under a structured cessation program with carbon monoxide breath testing. The investigators hypothesize that self-reported smoking status is underreported and that routine carbon monoxide breath testing will improve abstinence rates at the time of surgery.

DETAILED DESCRIPTION:
This study looks at patients who have been referred to our clinic for a potential hip and knee joint replacement surgery. Once it has been determined that the patient requires surgical replacement of either their hip or knee and is placed on our surgical waitlist, the patient will be asked if he or she would like to participate in the study. The investigators would ask all patients, both self-declared smokers and non-smokers, to participate. This study would include completing a smoking history questionnaire and a noninvasive carbon monoxide breath test. While smoking status is already assessed in the McGill University Health Centre preoperative questionnaire, the investigators intend on expanding these questions in study participants to better quantify their nicotine exposure.

ELIGIBILITY:
Inclusion Criteria:

* Adults ages 18-85 who require a primary total hip or knee replacement
* Any gender
* Smokers and non-smokers
* Osteoarthritis, rheumatoid arthritis, avascular necrosis

Exclusion Criteria:

* Patients who require revision surgery
* Previous fracture to affected area
* Emergency surgery
* Patients who do not understand, read or communicate in either French or English

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who have been referred to our outpatient orthopaedic clinic for a potential hip and knee joint replacement and have been placed on our surgical waitlist for surgery.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2021-02-18 (Actual); Primary Completion 2025-01-31 (Estimated); Study Completion 2025-01-31 (Estimated)

PRIMARY OUTCOMES:
True incidence of smokers among patients undergoing joint replacement | 15 minutes
  The percentage of subjects who declare themselves as smokers and non-smokers with elevated Co2 levels.

SECONDARY OUTCOMES:
To determine the incidence of patients who successfully quit smoking prior to surgery. | 20 minutes
  The percentage of subjects who were able to quit smoking under a structured cessation program with Carbon monoxide breath testing.

CONTACTS AND LOCATIONS:
Locations (1):
- Dr, Adam Hart, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No